CLINICAL TRIAL: NCT06831487
Title: Analysis of Line-Field Confocal Optical Coherence Tomography (LC-OCT) in the Characterization of Gingival Systemic Health, Gingivitis and Periodontitis and Effects of Periodontal Treatment
Brief Title: Analysis of Line-Field Confocal Optical Coherence Tomography (LC-OCT) in Characterization of Gingival Systemic Health, Gingivitis and Periodontitis
Acronym: Perio-LC-OCT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Associate Professor, University of Catania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-3307
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Gingival Diseases
Keywords: Periodontitis, gingivitis, LC-OCT
MeSH Terms: conditions — Gingival Diseases; Periodontitis; Gingivitis

STUDY DESIGN:
Intervention Model Description: Independently, patients with gingivitis, periodontitis and healthy patients will be evaluated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Analysis of Line-Field Confocal Optical Coherence Tomography (LC-OCT) in gingivitis (Active Comparator): Analysis of tissue changes pre and post non surgical periodontal treatment using Line-Field Confocal Optical Coherence Tomography (LC-OCT) in gingivitis patients
  Interventions: Device: Line-Field Confocal Optical Coherence Tomography (LC-OCT)
- Line-Field Confocal Optical Coherence Tomography (LC-OCT) periodontitis (Active Comparator): Line-Field Confocal Optical Coherence Tomography (LC-OCT) in periodontitis patients
  Interventions: Device: Line-Field Confocal Optical Coherence Tomography (LC-OCT)
- Line-Field Confocal Optical Coherence Tomography (LC-OCT) - Healthy patients (Placebo Comparator): Analysis of Line-Field Confocal Optical Coherence Tomography (LC-OCT) in healthy patients
  Interventions: Device: Line-Field Confocal Optical Coherence Tomography (LC-OCT)

INTERVENTIONS:
Device: Line-Field Confocal Optical Coherence Tomography (LC-OCT) — Analysis of Line-Field Confocal Optical Coherence Tomography (LC-OCT) in separate groups of patients with gingivitis, periodontitis and healthy patients
  Other Names: Line-Field Confocal Optical Coherence Tomography (LC-OCT) in all patients

SUMMARY:
The aim of the study is to identify tissue changes among healthy patients, patients with gingivitis and with periodontitis before and after treatment, by analyzing tissues changes through Line-Field Confocal Optical Coherence Tomography (LC-OCT)

DETAILED DESCRIPTION:
The tissue changes among healthy patients, patients with gingivitis and with periodontitis before and after treatment, by analyzing tissues changes through Line-Field Confocal Optical Coherence Tomography (LC-OCT) will be evaluated through changes on epithelium before and after non surgical periodontal treatment

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gingivitis or periodontitis by the presence of elevated bleeding or probing index or probing pocket depth

Exclusion Criteria:

* Smoking
* Any systemic diseases that could influence the gingival structure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual epithelial surface change | 6-months
  Analysis of disruption of superficial epithelium and basal line

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico G. Rodolico, Catania, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Study results